CLINICAL TRIAL: NCT00422799
Title: Phase II Study of Combination Bortezomib (Velcade PS-341) and Rituximab in Patients With Previously Untreated and Relapsed/Refractory Waldenstrom's Macroglobulinemia
Brief Title: Combination Bortezomib and Rituximab in Patients With Waldenstrom's Macroglobulinemia (WM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-008
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Results first posted 2018-01-26 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: relapsed Waldenstrom's macroglobulinemia; refractory Waldenstrom's macroglobulinemia; Velcade; WM
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Bortezomib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bortezomib and rituximab (Experimental): bortezomib and rituximab
  Interventions: Drug: Bortezomib; Drug: Rituximab

INTERVENTIONS:
Drug: Bortezomib — Once weekly for 3 weeks
  Other Names: Velcade
Drug: Rituximab — Intravenously once a week for the first and fourth weeks of a cycle
  Other Names: Rituxan

SUMMARY:
In this study, we are trying to find out if the combination of these two drugs is effective in treating Waldenstrom's macroglobulinemia (WM). The combination of these two drugs has not been studied for patients with relapsed or refractory macroglobulinemia. The U.S. Food and Drug Administration (FDA) has approved bortezomib for the treatment of multiple myeloma, a cancer that is closely related to Waldenstrom's macroglobulinemia.

DETAILED DESCRIPTION:
* Participants will receive 6 cycles of the study treatment with bortezomib and rituximab. Each cycle is 28 days long (4 weeks).
* Participants will receive Rituximab intravenously once a week for the first and fourth cycles only. Participants will receive bortezomib once a week for three weeks on and one week off every cycle, for a total of 6 cycles.
* During the rituximab infusion, the participants blood pressure and pulse will be monitored frequently. The rate of infusion may be decreased depending upon the side effects that are experienced.
* Blood samples will be collected before the first dose and on follow up with every cycle. Blood counts will also be performed every week.
* Routine physical exams will be performed at each evaluation. A PET/CAT scan of the chest, abdomen and pelvis at the end of treatment. This scan is required to assess the response of the participants disease.
* In order to learn more on how bortezomib and rituximab affect WM, a bone marrow biopsy will be performed.
* We anticipate that participants will complete the active therapy over a period of 6 cycles provided that they are benefiting from therapy and have not had any serious side effects. The participant will be followed every three months for 2 years for office visits and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients with previously untreated WM and those who have received prior therapy are eligible
* Must have received prior therapy for their WM and have relapsed or refractory WM.
* CD20 positive disease based on any previous bone marrow immuno-histochemistry or flow cytometric analysis performed up to 3 months prior to enrollment.
* Measurable disease
* ECOG Performance Status 0,1, or 2
* Total bilirubin < 2.0 mg/dl
* AST < 3 x ULN
* Life expectancy of greater than 12 weeks

Exclusion Criteria:

* Uncontrolled infection
* Other active malignancies
* Cytotoxic chemotherapy less than 3 weeks, or biologic therapy less than 2 weeks, or corticosteroids less than 2 weeks, prior to registration.
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational
* Known to be HIV positive or HEP B positive
* Radiation therapy less than 2 weeks prior to registration
* Grade 2 or greater peripheral neuropathy
* Myocardial infarction within 6 months rior to enrollment or has NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Hypersensitivity to bortezomib, boron, or mannitol
* Pregnant or breast feeding women
* Other investigational drugs within 14 days of enrollment
* Serious medical or psychiatric illness likely to interfere with participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-08-30 (Actual); Primary Completion 2015-10-09 (Actual); Study Completion 2015-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Result] Ghobrial IM, Hong F, Padmanabhan S, Badros A, Rourke M, Leduc R, Chuma S, Kunsman J, Warren D, Harris B, Sam A, Anderson KC, Richardson PG, Treon SP, Weller E, Matous J. Phase II trial of weekly bortezomib in combination with rituximab in relapsed or relapsed and refractory Waldenstrom macroglobulinemia. J Clin Oncol. 2010 Mar 10;28(8):1422-8. doi: 10.1200/JCO.2009.25.3237. Epub 2010 Feb 8. PMID 20142586

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bortezomib and Rituximab
Started | 63
Completed | 50
Not Completed | 13
Not completed — Withdrawal by Subject | 6
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 27
Age, Continuous [Median (Full Range); unit: years] | 63 [43 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 41
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate of Bortezomib and Rituximab (VR) in Patients With Relapsed or Refractory Waldenstrom's Macroglobulinemia (WM)
Description: Overall Response Rate= Minor response (>25%-50% reduction in monoclonal IgM from baseline + Partial Response (>50-90% reduction in monoclonal IgM from baseline)+ Complete Response (Disappearance of monoclonal protein by immunofixation; no histologic evidence of bone marrow involvement, resolution of any adenopathy/organomegaly (confirmed by CT scan), or signs or symptoms attributable to WM. Reconfirmation of the CR status is required at least 6 weeks apart with a second immunofixation.)
Time Frame: 2 Years
Population: Patients who had received at least one prior line of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 37
Participants | 30

2. Primary Outcome: Overall Response Rate of Bortezomib and Rituximab (VR) in Patients With Previously Untreated Waldenstrom's Macroglobulinemia (WM)
Description: as for outcome 1
Time Frame: 2 years
Population: Participants who were previously untreated.
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 26
Participants | 23

3. Secondary Outcome: Time to Progression in Patients With WM
Description: Time to progresion is the defined as the time from study entry to disease progression (PD) or death. Patients without PD are censored at the date of last disease evaluation. PD is defined as a greater than 25% increase in serum monoclonal IgM electrophoresis confirmed by a second measurement at least 2 weeks apart, or progression of clinically significant findings due to disease or symptoms attributable to WM.
Time Frame: 5 Years
Population: All enrolled participants.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 63
years | 1.6 [1.1 to 5]

4. Secondary Outcome: Duration of Response in Patients With WM
Description: Time from documentation of first response to progressive disease.
Time Frame: 5 Years
Population: All participants enrolled
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 63
years | 1.4 [0.6 to 5]

ADVERSE EVENTS:
Arm/Group | Bortezomib and Rituximab
All-Cause Mortality (participants affected / at risk) | 1/63
Serious Adverse Events (participants affected / at risk) | 11/63
Other Adverse Events (participants affected / at risk) | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib and Rituximab (N=63)
Infection (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib and Rituximab (N=63)
Edema limb (General disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Upper airway infection (Infections and infestations) | 4 (4)
Joint pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Muscle pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Allergic reaction (Immune system disorders) | 20 (20)
Dizziness (Nervous system disorders) | 7 (7)
Neuropathy-sensory (Nervous system disorders) | 32 (32)
ALT elevation (Investigations) | 6 (6)
AST elevation (Investigations) | 11 (11)
Alkaline phosphatase elevation (Investigations) | 7 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 28 (28)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 25 (25)
Nausea (Gastrointestinal disorders) | 25 (25)
Vomiting (Gastrointestinal disorders) | 9 (9)
Fatigue (General disorders) | 44 (44)
Fever without neutropenia (General disorders) | 6 (6)
Weight loss (Investigations) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 55 (55)
Leukopenia (Blood and lymphatic system disorders) | 36 (36)
Neutropenia (Blood and lymphatic system disorders) | 28 (28)
Thrombocytopenia (Blood and lymphatic system disorders) | 28 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less